CLINICAL TRIAL: NCT00085566
Title: A Phase I/II Trial to Assess the Tolerability of RAD 001 With Gefitinib in Patients With Glioblastoma Multiforme and Prostate Cancer and Efficacy in Patients With Castrate Metastatic Prostate Cancer
Brief Title: Everolimus and Gefitinib in Treating Patients With Progressive Glioblastoma Multiforme or Progressive Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-010; MSKCC-04010
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Brain and Central Nervous System Tumors; Prostate Cancer
Keywords: adult glioblastoma; recurrent prostate cancer; recurrent adult brain tumor; stage IV prostate cancer; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Prostatic Neoplasms; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — Everolimus; Gefitinib

ARMS (1):
- Everolimus (RAD-001) and Gefitinib (Experimental): •Phase I: Patients receive oral everolimus on day 1 and oral gefitinib once daily on days 8-21. Beginning on day 22, patients receive oral everolimus once weekly and oral gefitinib once daily. Treatment with the combination continues in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of everolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  •Phase II (prostate cancer patients only) (closed to accrual as of 10/19/2006): Patients receive oral everolimus (at the MTD determined in phase I) once weekly and oral gefitinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Drug: gefitinib

INTERVENTIONS:
Drug: everolimus
Drug: gefitinib

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by stopping blood flow to the tumor. Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining everolimus with gefitinib may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of everolimus when given together with gefitinib and to see how well they work in treating patients with progressive glioblastoma multiforme or (progressive metastatic prostate cancer closed to accrual 10/19/06).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of everolimus when given in combination with gefitinib in patients with progressive glioblastoma multiforme or (progressive castrate metastatic prostate cancer -closed to accrual as of 10/19/2006). (Phase I)
* Determine the safety and efficacy of this regimen in patients with progressive glioblastoma multiforme or (progressive castrate metastatic prostate cancer - closed to accrual as of 10/19/2006). (Phase II)

Secondary

* Determine whether a pharmacokinetic interaction exists between everolimus and gefitinib in patients treated with this regimen.
* Determine the association between clinical outcomes and markers that may predict sensitivity of a tumor in patients treated with this regimen.
* Determine the pharmacodynamic effects of this regimen on post-therapy tumor specimens and peripheral blood mononuclear cells from these patients.

OUTLINE: This is a phase I, open-label, non-randomized, dose-escalation study of everolimus followed by a phase II study.

* Phase I: Patients receive oral everolimus on day 1 and oral gefitinib once daily on days 8-21. Beginning on day 22, patients receive oral everolimus once weekly and oral gefitinib once daily. Treatment with the combination continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of everolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II (prostate cancer patients only) (closed to accrual as of 10/19/2006): Patients receive oral everolimus (at the MTD determined in phase I) once weekly and oral gefitinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Glioblastoma multiforme (GBM) (phase I only)

    * Progressive disease despite standard therapy
    * Progressive disease based on 1 of the following:

      * New or progressive (25% bidimensional increase) soft tissue masses on CT scan or MRI
      * New or prior lesions that have increased in size by physical examination
    * Patients who had prior interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true disease progression (rather than radiation necrosis) by positron-emission tomography scan, thallium scanning, magnetic resonance spectroscopy, or surgical documentation
  * Castrate metastatic prostate cancer (closed to accrual as of 10/19/2006) (phase I and II)

    * Progressive disease despite standard therapy AND castrate levels < 50 ng/dL of testosterone
    * Progressive disease based on 1 or more of the following:

      * A minimum of 3 rising levels of prostate-specific antigen (PSA) that are obtained 1 or more weeks apart OR 2 rising PSA values obtained more than 1 month apart with at least a 25% increase over the range of values
      * New or progressive (25% bidimensional increase) soft tissue masses on CT scan or MRI
      * New metastatic lesions
    * Patients on an antiandrogen as part of initial therapy must show disease progression after discontinuation of the antiandrogen
    * Patients who have not undergone surgical orchiectomy must continue with medical therapy (e.g., gonadotropin-releasing hormone analogs) to maintain castrate levels of serum testosterone
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3

Hepatic

* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine within 1.5 times ULN (< 1.95 mg/dL at MSKCC)

Cardiovascular

* No significant cardiovascular disease
* No congestive heart failure
* No New York Heart Association class III or IV cardiac disease
* No active angina pectoris
* No myocardial infarction within the past 6 months

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious medical illness
* No severe infection
* No severe malnutrition
* No other active malignancy except non-melanoma skin cancer

  * Patients are not considered to have an active malignancy if they have completed prior therapy and currently have a < 30% risk for relapse

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biological therapy
* No concurrent immunotherapy

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* Prior recent resection of recurrent or progressive GBM allowed provided patient has recovered
* More than 4 weeks since prior major surgery

Other

* Recovered from all prior therapy
* More than 4 weeks since prior investigational anticancer drugs
* No concurrent anticonvulsant that interacts with CYP3A4 (e.g., phenytoin, carbamazepine, or phenobarbital)
* No other concurrent cytotoxic therapy
* No other concurrent investigational or commercial agents or therapies for the malignancy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard I. Scher, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Neal Rosen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Lauren E. Abrey, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Vall d'Hebron University Hospital, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD 001 30 mg: 30 mg RAD 001 with Gefitinib in Patients with Glioblastoma Multiforme and Prostate Cancer
- RAD 001 50 mg: 50 mg RAD 001 with Gefitinib in Patients with Glioblastoma Multiforme and Prostate Cancer
- RAD 001 70 mg: 70 mg RAD 001 with Gefitinib in Patients with Glioblastoma Multiforme and Prostate Cancer
Period: Overall Study
Arm/Group | RAD 001 30 mg | RAD 001 50 mg | RAD 001 70 mg
Started | 3 | 3 | 57
Completed | 3 | 3 | 43
Not Completed | 0 | 0 | 14
Not completed — Adverse Event | 0 | 0 | 10
Not completed — Patient Not treated | 0 | 0 | 3
Not completed — Clinical progression | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAD 001 30 mg | RAD 001 50 mg | RAD 001 70 mg | Total
Number analyzed (Participants) | 3 | 3 | 57 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 32 | 34
  >=65 years | 2 | 2 | 25 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 11 | 11
  Male | 3 | 3 | 46 | 52

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Response will be evaluated in this study using the new international criteria Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | RAD 001 30 mg | RAD 001 50 mg | RAD 001 70 mg
Number analyzed (Participants) | 3 | 3 | 43
participants
  Partial Response (PR) | 0 | 0 | 2
  Stable Disease (SD) | 0 | 1 | 15
  Progression of Disease (POD) | 3 | 2 | 26

ADVERSE EVENTS:
Arm/Group | RAD 001 30 mg | RAD 001 50 mg | RAD 001 70 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 18/57
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 48/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD 001 30 mg (N=3) | RAD 001 50 mg (N=3) | RAD 001 70 mg (N=57)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ALT, SGPT (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac General, other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Death not associated w CTCAE term-Disease progression NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Extremity-lower (gait/walking) (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, Peritoneal cavity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infection, other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Mood alteration - Agitation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness - Extremity-lower (General disorders) | 0 (0) | 0 (0) | 1 (1)
Neurology - Other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pain - Head/headache (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Thrombosis/embolism (vascular access-related) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD 001 30 mg (N=3) | RAD 001 50 mg (N=3) | RAD 001 70 mg (N=57)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 8 (8)
ALT, SGPT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (8)
AST, SGOT (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (6)
Calcium, low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 10 (10)
Cholesterol, high (hypercholestremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Dyspnea (shortness of breath) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 8 (8)
Edema: limb (General disorders) | 0 (0) | 0 (0) | 5 (5)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 1 (1) | 12 (12)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 19 (19)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 20 (20)
Prothrombin Time and International Normalized Ratio (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 10 (10)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 17 (17)
Mucositis (Clincal exam)- Oral cavity (General disorders) | 0 (0) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4)
Partial Thromboplastin Time (PTT) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Pain - Bone (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Extremity-lower (gait/walking) (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes